CLINICAL TRIAL: NCT04165291
Title: Comparing a Fatherhood Focused Individual Intervention to Batterer Intervention to Reduce IPV and Child Maltreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000026789; 1R21HD099318-01A1 (NIH)
Record Dates: First submitted 2019-11-14; First posted 2019-11-15 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Intimate Partner Violence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F4C (Experimental): Participants randomized to the Fathers for Change (F4C) program.
  Interventions: Behavioral: F4C
- BIP (Active Comparator): Participants randomized to the Batterer Intervention Program (BIP).
  Interventions: Behavioral: BIP

INTERVENTIONS:
Behavioral: F4C — Fathers for Change (F4C) focuses on: 1) the fathering role to facilitate engagement, 2) RF to understand self, partner and children and emotion regulation skills to reduce IPV and child maltreatment. F4C focuses on understanding of emotional experiences, how they impact thinking and behaviors related to partners, co-parents and children. F4C clients will meet individually with their F4C therapist for 50 minutes per week over 16 weeks.
  Arms: F4C
Behavioral: BIP — The Batterer Intervention Program (BIP) is a psychoeducational intervention that will be delivered in 50- minute individual weekly sessions over 16 weeks. The intervention focuses on the impact of violence on victims, power and control tactics, and societal influences supporting men's violence toward women. The intervention includes didactics and experiential exercises including role plays to teach anger management skills.
  Arms: BIP

SUMMARY:
This randomized trial will test a newly developed intervention aimed at fathers who have a history of family violence compared to a standard batterer intervention program.

DETAILED DESCRIPTION:
This study will expand on Fathers for Change (F4C), a novel intervention for fathers with histories of perpetrating intimate partner violence (IPV). F4C is designed to meet a significant unmet intervention need for fathers who have a history of family violence who are not helped by currently available batterer intervention programs (BIPs). BIPs that are currently available nationally have shown limited efficacy with high rates of repeat violence.

This project will provide needed data to further develop F4C and move to a Stage II efficacy trial by: 1) revising the BIP group intervention manual to be delivered in an individual treatment format; 2) develop a fidelity measure for F4C and the BIP; 4) conduct a stage 1b randomized trial (consistent with the stage model of intervention development) to show initial feasibility, acceptability and intervention signal with the targeted population.

Sixty fathers with a history of IPV who have already failed a treatment as usual group BIP will be randomly assigned to F4C or an individually delivered comparable dose of BIP. Reflective functioning and emotion regulation will be examined as the mechanisms through which Fathers for Change reduces IPV and child maltreatment risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* A reported an incident of IPV (pushing, slapping, kicking) within the last 12 months prior to screening (based on court/police records, partner or self- report);
* have at least one biological child aged 6 months to 7 years with whom they have contact in person or by phone/facetime etc. at least monthly;
* are able to complete assessments in English;
* agree to have their female coparents (mother of the youngest child) contacted as collateral informants and for consent for participation of their shared child.

Exclusion Criteria:

* Men who have an active full/no contact protective order pertaining to their child since this will preclude participation in the father-child play assessment (many men will have full no-contact orders with their partners, but it is more common for men to still be allowed at least supervised contact with their children even with a full/no contact order with their partner);
* physiological addiction to a substance that requires detoxification. Fathers will be evaluated using the Addiction Severity Index and urine toxicology screens. If fathers report difficulties with physiological withdrawal from substances (e.g. delirium tremens, shaking, nausea) they will be referred for detox services. They can be re-evaluated following a detox program with documentation from the detox center of successful completion and clean urine screen.;
* anyone with a cognitive impairment that will not allow for understanding of the study interventions (a mini mental state score <25);
* anyone with a current untreated psychotic disorder;
* anyone currently suicidal or homicidal based on screening using the BSI.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla Stover, PhD, Principal Investigator — Associate Professor at the Yale University School of Medicine Child Study Center
Locations (1):
- Carla Stover, Hamden, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fathers for Change: Participants randomized to the Fathers for Change (F4C) program.
  F4C: Fathers for Change (F4C) focuses on: 1) the fathering role to facilitate engagement, 2) RF to understand self, partner and children and emotion regulation skills to reduce IPV and child maltreatment. F4C focuses on understanding of emotional experiences, how they impact thinking and behaviors related to partners, co-parents and children. F4C clients will meet individually with their F4C therapist for 50 minutes per week over 18 weeks.
- Duluth Domestic Violence Program (BIP): Participants randomized to the Batterer Intervention Program (BIP).
  BIP: The Batterer Intervention Program (BIP) is a psychoeducational intervention that will be delivered in 50- minute individual weekly sessions over 18 weeks. The intervention focuses on the impact of violence on victims, power and control tactics, and societal influences supporting men's violence toward women. The intervention includes didactics and experiential exercises including role plays to teach anger management skills.
Period: Overall Study
Arm/Group | Fathers for Change | Duluth Domestic Violence Program (BIP)
Started | 30 | 30
Completed | 20 | 21
Not Completed | 10 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fathers for Change | Duluth Domestic Violence Program (BIP) | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (7.7) | 30.6 (7.4) | 33.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 30 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 17 | 32
  White | 4 | 3 | 7
  More than one race | 6 | 9 | 15
  Unknown or Not Reported | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Completion Rate
Description: To test the hypothesis that fathers randomized to F4C will have higher completion rates than those in the individual BIP treatment, chi-square analysis will be used to examine between group differences in treatment completion.
Time Frame: 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Fathers for Change | Duluth Domestic Violence Program (BIP)
Number analyzed (Participants) | 30 | 30
Participants | 20 | 21

2. Primary Outcome: Working Alliance Inventory Sum Score
Description: To test the hypothesis that fathers randomized to F4C will report greater overall working alliance, analysis of variance will be used to test between group difference in overall working alliance between F4C and BIP at week 8 of intervention (approximately mid-point). The Working Alliance Inventory (WAI-therapist version) will be used to measure working alliance among clinicians and clients. The WAI for therapists measures the strength of the working alliance with the client with 36 items utilizing a 5-point Likert scale. The minimum score is 0, the maximum score is 180. Higher sum score indicates a stronger working alliance.
Time Frame: 8 weeks
Population: Working Alliance was measured at 8 weeks from start of the interventions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fathers for Change | Duluth Domestic Violence Program (BIP)
Number analyzed (Participants) | 25 | 23
score on a scale | 62.52 (8.96) | 55.82 (6.77)
Statistical Analysis 1: Comparison: Fathers for Change vs Duluth Domestic Violence Program (BIP); Test type: Superiority; p < .01, ANOVA

3. Primary Outcome: Client Satisfaction Sum Score
Description: To test the hypothesis that fathers randomized to F4C will report greater overall satisfaction, analysis of variance will be used to test between group difference in overall client satisfaction between F4C and BIP. Satisfaction scores range from 2 to 8 with 8 indicating greater overall satisfaction with the services received.
Time Frame: 18 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fathers for Change | Duluth Domestic Violence Program (BIP)
Number analyzed (Participants) | 24 | 18
score on a scale | 7.75 (.68) | 7.33 (.84)
Statistical Analysis 1: Comparison: Fathers for Change vs Duluth Domestic Violence Program (BIP); Test type: Other; p = .08, ANOVA

4. Secondary Outcome: Reflective Functioning
Description: Reflective functioning will be assessed using the Parent Development Interview-Revised (PDI). The PDI is a 40-item semi-structured interview that assesses reflective functioning through questions about child-rearing and the ways respondents are like or unlike their own parents. Interviews will be audio recorded and transcribed verbatim for scoring. Interviews are coded on a scale of 1 to 9 with 1 being poor and 9 being excellent reflective functioning. A score of 3 or less is considered very poor.
Time Frame: Baseline and 18 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Fathers for Change | Duluth Domestic Violence Program (BIP)
Number analyzed (Participants) | 22 | 20
score on a scale
  Baseline | 2.46 (.157) | 2.57 (.165)
  Posttreatment | 2.39 (.121) | 2.23 (.127)
Statistical Analysis 1: Comparison: Fathers for Change vs Duluth Domestic Violence Program (BIP); Test type: Superiority; p = .116, Repeated Measures Analysis of Variance

5. Secondary Outcome: Emotional Regulation
Description: Emotional regulation will be assessed with the Difficulties in Emotion Regulation Scale-short form (DERS-SF). The DERS-SF is an 18-item self-report measure scored on a 5-point Likert-type scale where higher scores indicate greater difficulty in emotional regulation. Scores range from 18-90.
Time Frame: Baseline and 18 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Fathers for Change | Duluth Domestic Violence Program (BIP)
Number analyzed (Participants) | 22 | 21
score on a scale
  Baseline | 34.61 (2.07) | 28.64 (2.12)
  Post-Treatment | 29.20 (1.71) | 28.32 (1.76)
Statistical Analysis 1: Comparison: Fathers for Change vs Duluth Domestic Violence Program (BIP); Test type: Superiority; p < .05, Mixed Models Analysis; Mean Difference (Final Values) = 5.146

6. Secondary Outcome: Intimate Partner Violence
Description: The TimeLine Follow-back-Spousal Violence will be used to characterize the frequency of intimate partner violence.
Time Frame: 18 weeks
Population: imputation for missing data across weeks to increase sample size.
Measure: Mean (Standard Deviation); unit: Events/weeks
Arm/Group | Fathers for Change | Duluth Domestic Violence Program (BIP)
Number analyzed (Participants) | 27 | 25
Events/weeks | 1.70 (4.57) | 4.28 (7.41)
Statistical Analysis 1: Comparison: Fathers for Change vs Duluth Domestic Violence Program (BIP); Test type: Superiority; p = .13, ANOVA

7. Secondary Outcome: Child Maltreatment
Description: Child maltreatment risk will be assessed using TimeLine Follow-back to assess the frequency of behaviors characterized as child maltreatment.
Time Frame: 18 weeks
Measure: Mean (Standard Deviation); unit: Events/weeks
Arm/Group | Fathers for Change | Duluth Domestic Violence Program (BIP)
Number analyzed (Participants) | 27 | 25
Events/weeks | 1.19 (2.47) | 3.48 (12.50)
Statistical Analysis 1: Comparison: Fathers for Change vs Duluth Domestic Violence Program (BIP); Test type: Superiority; p = .35, ANOVA

ADVERSE EVENTS:
Time Frame: 19 weeks
Description: In our study we included arrest/incarceration as serious adverse events given the nature of our population with significant criminal histories.
Arm/Group | Fathers for Change | Duluth Domestic Violence Program (BIP)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 3/30 | 1/30
Other Adverse Events (participants affected / at risk) | 3/30 | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fathers for Change (N=30) | Duluth Domestic Violence Program (BIP) (N=30)
Arrest and Incarceration (Social circumstances) | 3 (4) | 1 (1) — Arrest and incarceration for intimate partner violence or drug related charges
Hospitalization (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Father was hit by a car
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fathers for Change (N=30) | Duluth Domestic Violence Program (BIP) (N=30)
ER Visits (General disorders) | 1 (2) | 1 (1) — Participant visits emergency department for injury or illness
Car Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
COVID diagnosis (General disorders) | 1 (1) | 0 (0) — Participant Tested positive for COVID had not visited the clinic in person

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT04165291/Prot_SAP_000.pdf